CLINICAL TRIAL: NCT01822730
Title: A Multiple-Center, Randomized, Double-Blind Study of Comparison of Paliperidone and Risperidone for Treatment of Patirnts With Methamphetamine-Associated Psychosis
Brief Title: A Comparison of Paliperidone and Risperidone for Treatment of Patirnts With Methamphetamine-Associated Psychosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wei Hao (Other)
Responsible Party: Sponsor-Investigator, Wei Hao, The Second Xiangya Hospital of Cental South University, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100000-068943
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine-Associated Psychosis; Aripiprazole; Risperidone
MeSH Terms: interventions — Paliperidone Palmitate; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paliperidone (Experimental): paliperidone arm,6mg/pill,6-12mg/day,non-forced titration method.last2-4weeks.
  Interventions: Drug: paliperidone
- .Risperidone (Active Comparator): Risperidone arm and placebo tables,1mg/pill,2mg-6mg/day,non-forced titration method.last2-4weeks
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: paliperidone — Paliperidone group,6mg/pill,6mg-12mg/day non-forced titration method,last 2-4weeks
  Other Names: Paliperidone Extended-Release Tablets; Invega
  Arms: paliperidone
Drug: Risperidone — Risperidone group,1mg/pill,2mg-6mg/day non-forced titration method,last 2-4weeks
  Other Names: Risperdal H20070057
  Arms: .Risperidone

SUMMARY:
Methamphetamine-associated psychosis (MAP) has been considered a pharmacological or environmental pathogen model of schizophrenia (SCZ) due in part to similarities in clinical presentation (i.e. paranoia, hallucinations, disorganized speech, and negative symptoms), response to treatment (e.g.neuroleptics),and pathologic mechanisms (e.g. central dopaminergic neurotransmission) of both conditions. Both paliperidone and risperidone are second generation antipsychotics，but have same pharmacological effects of antipsychotic treatment and paliperidone may have more efficacy and safty.This study was designed to examine the acute efficacy, safety, and tolerability of paliperidone and risperidone for patients with MAP.

DETAILED DESCRIPTION:
Methods:A Multiple-Center, Randomized, Double-Blind.

ELIGIBILITY:
Inclusion Criteria:

1. Patients,Diagnostic and Statistical Manual of Mental Disorders 4thed. (DSM-IV) criteria for Methamphetamine-Associated Psychosis.
2. Must sign a Information consent form.
3. Required to provide detailed address and phone number

Exclusion Criteria:

1. Serious organic disease.
2. Suicide ideation or hurt others.
3. Taking antipsychotic within two weeks before.
4. drug allergy to Risperidone or paliperidone.
5. pregnancy and breastfeeding women.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The severity of psychosis | up to 4 weeks. participants will be followed for the duration of hospital stay
  Positive and Negative Syndrome Scale

SECONDARY OUTCOMES:
Clinical general status | up to 4 weeks. participants will be followed for the duration of hospital stay
  Clinical general rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hao, MD., Ph.D., Study Director — Central South University
Locations (1):
- The Second Xiangya Hospital of Central University, Changsha, Hunan, China

REFERENCES:
- [Derived] Wang G, Ding F, Chawarski MC, Hao W, Liu X, Deng Q, Ouyang X. Randomized Controlled Trial of Paliperidone Extended Release Versus Risperidone for the Treatment of Methamphetamine-Associated Psychosis in Chinese Patients. Front Psychiatry. 2020 Apr 1;11:237. doi: 10.3389/fpsyt.2020.00237. eCollection 2020. PMID 32296355